CLINICAL TRIAL: NCT00062166
Title: Evaluation of the Natural History and Management of Pancreatic Lesions Associated With Von Hippel-Lindau
Brief Title: Natural History and Management of Pancreatic Lesions in Von Hippel-Lindau Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030145; 03-C-0145; NCT01444950 (obsolete NCT alias)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Von Hippel-Lindau Disease
Keywords: Imaging Studies; Rate of Tumor Growth; Familial Cancer Syndrome; Surgical Resection
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Von Hippel-Lindau disease (VHL) is an inherited cancer syndrome. Patients are at risk for developing pancreatic cysts and tumors. These tumors are more aggressive in some people than in others. To learn more about this disease, its genetic cause and how best to treat it, this study will 1) identify patients with VHL who have pancreatic lesions; 2) examine the characteristics of the lesions and how fast they grow; 3) study how well imaging tests can reveal lesion characteristics that will help in diagnosis; and 4) perform genetic studies using blood and, when possible, tissue samples.

Patients 12 years of age and older with VHL involving the pancreas may be eligible for this study. Participants will undergo some or all of the following tests and procedures:

* Interviews with a cancer doctor, cancer nurses, and a surgeon (if surgery is recommended).
* Computed tomography (CT) scan of the abdomen, chest, or pelvis. This test uses x-rays to produce images of body tissues and organs in small sections.
* Magnetic resonance imaging (MRI) of the abdomen. This test uses radio waves and a strong magnetic field to produce images of body tissues and organs.
* Ultrasound of the abdomen. This test uses sound waves to create images body tissues and organs.
* Blood tests for routine laboratory chemistries, for tests specific to the pancreas, and for genetic studies
* 24-hour urine studies

After the tests are completed, the doctor will discuss the results with the patient. Patients with a pancreatic tumor that requires surgery will be offered the option of an operation to remove as much tumor as possible. Patients with lesions that are not appropriate for surgery will be asked to return to National Institutes of Health (NIH) for scans and x-rays every year to monitor growth of the lesions. If surgery should become advisable in the future, the option will be discussed at that time. Patients with pancreatic cysts will be asked to return to NIH every 2 years for scans and x-rays to monitor their condition.

DETAILED DESCRIPTION:
Background:

Patients with the familial cancer syndrome von Hippel-Lindau (VHL) demonstrate manifestations in a variety of organs among them the pancreas. Pancreatic manifestations can range from benign cysts and micro cystic adenomas to neuroendocrine tumors of the pancreas which are capable of regional and distant spread. These neuroendocrine tumors can result in life-threatening complications.

This protocol is designed to identify VHL patients with pancreatic manifestations and to follow these patients with serial imaging studies and germ line and tissue genetic analysis.

Objectives:

To identify patients with VHL having pancreatic lesions defined by simple cysts, microcystic adenomas, neuroendocrine tumors and other solid lesions of the pancreas.

To follow patients with VHL and pancreatic manifestations by serial examination with non-invasive imaging studies.

For patients with solid lesions of the pancreas, to determine the rate of growth and to correlate the growth rate with clinical measures of disease progression.

To validate non-invasive imaging methods for differentiating benign solid lesions from lesions with malignant potential.

To characterize the time from initial presentation with pancreatic tumors to the time that surgery is recommended.

Eligibility:

Patients greater than or equal to 12 years of age who have been diagnosed with VHL.

Patients/parent must be able to sign an informed consent and be willing to return to National Institutes of Health (NIH) for follow-up.

Design:

Demographic data will be collected from the medical record and patient interview for each patient participant. Data will be securely stored in a computerized database.

Patients will be evaluated by the Urologic Oncology Branch personnel as indicated to rule out or manage other manifestations of VHL. Imaging studies of regions other than the chest and abdomen will be dictated by best clinical practice for the workup and management of VHL manifestations as has been previously published.

All patients enrolled on this study will be offered genetic counseling by a trained genetic counselor.

After their initial on-study evaluation, patients who are not found to have solid lesions of the pancreas but rather have only cystic disease of the pancreas, will be re-screened every two years with non-invasive imaging studies.

Surgical resection of solid lesions of the pancreas will be recommended based on previously published criteria.

Based on our analysis of likelihood of tumor growth or risk of metastasis, data will be analyzed every two years and appropriate revisions will be made to the surgical management guidelines, if indicated by data analysis.

Projected accrual will be 25 patients per year for a total of 15 years. Thus, we anticipate accruing 600 patients on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who have been diagnosed with Von Hippel Lindau (VHL) using the following criteria: either germ line analysis (12) or clinical criteria and a family history (8, 12) and who have at least 1 pancreatic manifestation of VHL as documented on any non-invasive imaging study. These manifestations include:

1. Pancreatic cyst(s).
2. Solid lesions suspicious for microcystic adenoma(s).
3. Solid enhancing lesions suspicious for primitive neuroectodermal tumor (PNET)(s).
4. Any other solid lesion(s) of the pancreas.

Age greater than or equal to 12 years of age.

Patients must be willing to return to National Institutes of Health (NIH) for follow-up.

Patients/parent must be able to sign an informed consent.

EXCLUSION CRITERIA:

Patients unwilling to undergo serial non-invasive imaging.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Von Hippel-Lindau (VHL) disease. Von Hippel-Lindau (VHL) is an inherited cancer syndrome. Patients are at risk for developing pancreatic cysts and tumors. Other tumors include kidney cancers, pheochromocytoma, eye and central nervous system tumors. These tumors occur at a higher frequency rate than normal population.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2003-04-11 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clifford SC, Maher ER. Von Hippel-Lindau disease: clinical and molecular perspectives. Adv Cancer Res. 2001;82:85-105. doi: 10.1016/s0065-230x(01)82003-0. PMID 11447766
- [Background] Glenn GM, Daniel LN, Choyke P, Linehan WM, Oldfield E, Gorin MB, Hosoe S, Latif F, Weiss G, Walther M, et al. Von Hippel-Lindau (VHL) disease: distinct phenotypes suggest more than one mutant allele at the VHL locus. Hum Genet. 1991 Jun;87(2):207-10. doi: 10.1007/BF00204184. PMID 2066108
- [Background] Gnarra JR, Duan DR, Weng Y, Humphrey JS, Chen DY, Lee S, Pause A, Dudley CF, Latif F, Kuzmin I, Schmidt L, Duh FM, Stackhouse T, Chen F, Kishida T, Wei MH, Lerman MI, Zbar B, Klausner RD, Linehan WM. Molecular cloning of the von Hippel-Lindau tumor suppressor gene and its role in renal carcinoma. Biochim Biophys Acta. 1996 Mar 18;1242(3):201-10. doi: 10.1016/0304-419x(95)00012-5. No abstract available. PMID 8603073

RESULTS

PARTICIPANT FLOW:
Groups:
- Von Hippel Lindau: Von Hippel-Lindau disease (VHL) is an inherited cancer syndrome. Patients are at risk for developing pancreatic cysts and tumors. Other tumors include kidney cancers, pheochromocytoma, eye and central nervous system tumors. These tumors occur at a higher frequency rate than normal population.
Period: Overall Study
Arm/Group | Von Hippel Lindau
Started | 340
Completed | 334
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 327
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 310
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 15
  White | 287
  More than one race | 1
  Unknown or Not Reported | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 340

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pancreatic Lesions Defined by Simple Cysts, Microcystic Adenomas, Neuroendocrine Tumors & Other Solid Lesions of the Pancreas Who Had Significant Growth in Lesions or Symptoms Related to the Lesions Requiring Surgical Intervention
Description: Pancreatic lesions defined by simple cysts, microcystic adenomas, neuroendocrine tumors and other solid lesions of the pancreas were evaluated by 18F Fludeoxyglucose (18F-FDG-PET) imaging to determine if the participant developed metastatic disease (e.g. tumor spreads to different organs).
Time Frame: 8 years
Population: Only 319/340 records are available in the database program for this outcome measure. No records are available for the remaining 21 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 319
Participants | 47

2. Secondary Outcome: Percentage of Participants With Exon 3 Mutation Compared to Participants With Exon 1 or 2 Von Hippel Lindau (VHL) Mutations Who Required an Intervention
Description: Percentage of patients by the location of germline VHL mutations.
Time Frame: 8 years
Population: The exon mutation information only is available in 63 patients. This protocol did not repeat the gene testing in any of the patients.
Measure: Number; unit: percentage of participants
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 63
percentage of participants
  exon 1 and 2 mutation | 53.97
  exon 3 mutation | 46.03
Statistical Analysis 1: Comparison: Von Hippel Lindau; Test type: Non-Inferiority — Time dependent risk for requiring an intervention for pancreatic neuroendocrine tumors (PNET), among 63 patients with PNETs with diameter >1.2 and <3 cm, and a known position of germline VHL pathogenic variant (n=63). Comparison between exon 3 vs exon 1 and 2; p = 0.02, Regression, Cox; Hazard Ratio (HR) = 3.3, 95% CI 2-sided [1.2 to 9.1]

3. Secondary Outcome: Number of Participants From Which We Obtained Tissue From Pancreatic Lesions and Normal Tissue for Genetic Analysis
Description: Count of participants from which we obtained tissue from pancreatic tumor and normal tissue (when applicable) for Deoxyribonucleic acid (DNA), ribonucleic acid (RNA), and proteins extraction.
Time Frame: initiation of study therapy until 2009, approximately 6 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 319
Participants | 46

4. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Groups:
- Von Hippel Lindau: Von Hippel-Lindau disease (VHL) is an inherited cancer syndrome. Patients are at risk for developing pancreatic cysts and tumors. These tumors are Von Hippel-Lindau disease (VHL) is an inherited cancer syndrome. Patients are at risk for developing pancreatic cysts and tumors. Other tumors include kidney cancers, pheochromocytoma, eye and central nervous system tumors. These tumors occur at a higher frequency rate than normal population.
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 340
Participants | 22

5. Secondary Outcome: Number of Participants With Missense or Non-missense Mutations
Description: Count of participants by the type of Von Hippel-Lindau (VHL) gene mutations.
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Von Hippel Lindau
Number analyzed (Participants) | 156
Participants
  missense mutations | 76
  non-missense mutations | 80

ADVERSE EVENTS:
Time Frame: 8 years
Description: Because this is natural history protocol, deaths or complications from treatments were not considered as AE or SAE. However, because 22 deaths are noted in the mortality module, 22 deaths are also noted in the SAEs per the Results Data Elements Definitions which state that "SAEs include AEs that result in death. Typically, the event(s) leading to death is listed as an AE Term in the SAE table and the number of participants who died due to any cause are reported in the All-Cause Mortality table."
Arm/Group | Von Hippel Lindau
All-Cause Mortality (participants affected / at risk) | 22/340
Serious Adverse Events (participants affected / at risk) | 22/340
Other Adverse Events (participants affected / at risk) | 0/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Von Hippel Lindau (N=340)
Death (General disorders) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT00062166/Prot_SAP_ICF_000.pdf